CLINICAL TRIAL: NCT04138095
Title: Virtual Reality as an Adjunct to Management of Pain and Anxiety in Palliative Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riverview Health Centre (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other); Riverview Health Centre Foundation (Other)
Responsible Party: Principal Investigator, Stefan Riel, Family Physician and Palliative Care Fellow, Riverview Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RiverviewHC
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Cancer; Heart Failure; Copd; ALS
Keywords: Palliative Care; Virtual Reality; Pain; Anxiety
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Within subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality (Other): As this is a within subject design, participants will act as their own control. Participants will have access to their baseline opioids and benzodiazepines for pain and anxiety. Every second day they will have access to virtual reality as an adjunct to their opioids and benzodiazepines to manage their symptoms
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Participants will have access to an Oculus Quest Virtual Reality Headset every second day as an alternative to opioids for pain management and benzodiazepines for anxiety management

SUMMARY:
Virtual reality has been shown to be an effective way to treat pain and anxiety in various different settings. Palliative care is an area of medicine that often deals with patients suffering from pain and anxiety. The medication used to manage these symptoms are often opioids and benzodiazepines due to their rapid onset however they do have a significant side effect burden on patients. Very few studies have looked at the effect of virtual reality in this patient population. The goal of this study is to measure if virtual reality can decrease the required amount of medication used in managing pain and anxiety in palliative care. The secondary outcome will look at perceived benefit by patients

DETAILED DESCRIPTION:
Virtual reality has been available for many years and is starting to gain traction in clinical setting in varied fields with multiple applications. Some of the primary clinical settings that virtual reality has shown benefit are in pain attenuation and mental health, particularly anxiety. Palliative Care is a field of medicine that most patients have both pain and anxiety to a certain degree. The medications used to manage this (opioids, benzodiazepines) are used but not without side effects to the patient as well as cost to the medical system. So far, there are very few studies looking at the effect of virtual reality on symptom burden in palliative care. The primary outcome of this study would be to look at virtual reality's role in decreasing breakthrough opioids use for pain and benzodiazepine use for anxiety by decreasing symptoms experienced by patients by providing them with an immersive computer generated experience. The secondary outcome of this study will be patient's perception of symptoms with the use of virtual reality.

Virtual reality has been shown to be effective in many areas of medicine, particularly in pain management and mental health. Studies utilizing VR in pain management have commonly been done with burn victims, as burns are thought to be among the most painful injuries people sustain. Using a within subject design where the patient is his/her own control, these studies have shown an observable benefit in decreasing pain as well as cutting down on the opioid doses required to get analgesia in patients requiring wound debridement and physiotherapy in both adults and children. The investigator's patient population in palliative care is susceptible to painful metastases, pressure ulcers, and other causes of pain, which are comparable to pain experienced by burn victims. Therefore, the results of theses studies are relevant and may prove beneficial for patients receiving palliative care.

In this study, patients will receive alternating days of standard palliative care and standard palliative care with virtual reality as an option for symptom management for a total of 4-10 days. Patients will be randomized to start with standard care with virtual reality or start with standard care alone. The immersive virtual reality experience would be delivered through an Oculus Quest. There will be 3 different software options that can be used based on preference. Patients will be asked the degree of pain/anxiety prior to applying the virtual reality headset and then the same scale immediately after indicating their pain/anxiety during the experience. After the 4-10 days, breakthrough use of opioids and benzodiazepines during days with standard care and virtual reality will be compared to breakthrough use with standard care alone.

It is anticipated that the use of virtual reality will decrease the amount of medication necessary to manage symptoms of pain and/or anxiety. It is also anticipated that this will provide the patient with a pleasant respite from their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled on the palliative care program and admitted to Riverview Health Centre Palliative Care unit
* Using 2 or more doses above their regular scheduled dose of opioids and/or benzodiazepines
* Reading/understanding fluency in English

Exclusion Criteria:

* Patients who cannot wear the headset due to a structural cause (i.e. head and neck malignancy making wearing headset uncomfortable
* Patients who are legally blind
* Participants who cannot tolerate the HMD and VR due to simulator sickness will have to be withdrawn from the study by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Opioid and Benzodiazepine use | 10 days
  Number of additional doses of opioids and benzodiazepines used on standard of care days will be compared to additional doses of opioids and benzodiazepines used on standard of care and virtual reality days

SECONDARY OUTCOMES:
Patient perception of benefit | 10 days
  Patient will be asked to complete a Visual Analogue Scale for pain (scale from 0 to 10, 0 being no pain and 10 being worse pain imaginable) and and/or Visual Analogue Scale for anxiety (scale from 0 to 10, 0 being no anxiety/calm and 10 being extremely anxious/fearful) immediately prior to virtual reality use and immediately after use. The two values will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riel, MD, Principal Investigator — University of Manitoba Palliative Care Program
Locations (1):
- Riverview Health Centre, Winnipeg, Manitoba, Canada